CLINICAL TRIAL: NCT00479050
Title: Phase 1 Study of Combination Chemoembolization and Radiofrequency Ablation for Hepatocellular Carcinoma Greater Than 3 cm
Brief Title: Combination Chemoembolization and Radiofrequency Ablation for Hepatocellular Carcinoma Greater Than 3 cm
Acronym: TACE-RFA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2001HCC; 03BS035
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma,treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: chemoembolization ,Radiofrequency ablation

SUMMARY:
Combined the chemoembolization and Radiofrequency ablation for the hepatocellular carcinoma greater than 3 cm,the ablation volume of coagulation necrosis can be significantly increased,which may be enable effective treatment of patients with HCC greater than 3 cm.

DETAILED DESCRIPTION:
To assess whether the effectiveness of a combination of transcatheter arterial chemoembolization(TACE) and radiofrequency ablation(RFA) is superior to TACE and RFA alone in treatment of patients with hepatocellular carcinoma(HCC)greater than 3 cm and to analyze the factors affecting the outcomes.

The patients with HCC of 3 or fewer lesions, each 3cm greater in diameter entered this randomized controlled trial. The primary end point was survival, and the secondary end points were tumor response.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria were:

1. Not indicated for resection,
2. Liver function of Child-Pugh class A or B,
3. 3 or fewer lesion, each 3 cm greater and 7.5 cm less in greatest diameter,
4. No portal vein involvement or extrahepatic metastasis,
5. Lesions located at least 5mm away from the hepatic hilum or gall bladder and the common bile duct,
6. Platelet count≥6.0×103/mm3 and the prothrombin activity≥60%, and
7. No previous HCC treatment.

Exclusion Criteria:

Exclusion criteria were:

1. Encephalopathy,
2. Refractory ascites,
3. Active gastrointestinal bleeding,
4. Renal failure.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2001-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years

SECONDARY OUTCOMES:
tumor response | 1-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang Qi Liang, MD,PhD, Study Chair — Dept. of Radiology

REFERENCES:
- [Derived] Cheng BQ, Jia CQ, Liu CT, Fan W, Wang QL, Zhang ZL, Yi CH. Chemoembolization combined with radiofrequency ablation for patients with hepatocellular carcinoma larger than 3 cm: a randomized controlled trial. JAMA. 2008 Apr 9;299(14):1669-77. doi: 10.1001/jama.299.14.1669. PMID 18398079 (Retraction: PMID 19380477 DeAngelis CD, Fontanarosa PB. JAMA. 2009 May 13;301(18):1931)